CLINICAL TRIAL: NCT07398261
Title: Efficacy of Mirabegron for Treatment of Non-monosymptomatic Nocturnal Enuresis in Children
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Menoufia University (Other)
Responsible Party: Principal Investigator, Mohammed Ali abdelghaffar, Assistant lecturer of urology, Menoufia University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Urol9/2023
Record Dates: First submitted 2023-08-29; First posted 2026-02-09 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Treatment of Non-monosymptomatic Nocturnal Enuresis
MeSH Terms: interventions — mirabegron; N-(4-((5-(hydroxy(phenyl)methyl)pyrrolidin-2-yl)methyl)phenyl)-4-oxo-4,6,7,8-tetrahydropyrrolo(1,2-a)pyrimidine-6-carboxamide

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Mirabegron 25 mg (Active Comparator): Patients received mirabegron 25 mg orally
  Interventions: Drug: Mirabegron 25 MG
- no intervention (No Intervention): no intervention

INTERVENTIONS:
Drug: Mirabegron 25 MG — Evaluate the efficacy of individual mirabegron or in combination for treatment of non-monosymptomatic nocturnal enuresis in children
  Other Names: vibegron
  Arms: Mirabegron 25 mg

SUMMARY:
This phase 3 clinical trial will compare use of individual treatment with mirabegron or desmopressin and their combination for treatment of non-monosymptomatic nocturnal enuresis in children

ELIGIBILITY:
Inclusion Criteria:

- Non-monosymptomatic nocturnal enuresis

Exclusion Criteria:

* monosymptomatic nocturnal enuresis

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 151 (Estimated)
Dates: Start 2023-08-28 (Actual); Primary Completion 2026-09-01 (Estimated); Study Completion 2026-11-01 (Estimated)

PRIMARY OUTCOMES:
Partial or complete response | 18 months

CONTACTS AND LOCATIONS:
Locations (1):
- Menoufia faculty of medicine, Shibīn al Kawm, Monufia Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol (2024-12-11): https://cdn.clinicaltrials.gov/large-docs/61/NCT07398261/Prot_000.pdf